CLINICAL TRIAL: NCT05722925
Title: Prospective Study Evaluating the Role of Axumin® (Fluciclovine or 18F-FACBC) PET in Patients With Biochemical Recurrence of Prostate Cancer and a Negative PSMA PET
Brief Title: Evaluating Fluciclovine PET in Patients With Biochemical Recurrence of Prostate Cancer and a Negative PSMA PET
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Blue Earth Diagnostics (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Nadine Mallak, MD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00024659
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fluciclovine PET/CT (Experimental): Participants will undergo Fluciclovine PET/CT within 30 days of a negative or equivocal PSMA PET scan. After the Fluciclovine PET/CT, the patient will follow up with their treating physician as per standard-of-care. The research team will collect clinical and imaging data at 6 months post Fluciclovine-PET/CT.
  Interventions: Drug: Fluciclovine PET/CT

INTERVENTIONS:
Drug: Fluciclovine PET/CT — 8 mCi (± 20%) of Fluciclovine administered as a bolus intravenous injection
  Other Names: 18F-FACBC; Axumin®

SUMMARY:
The purpose of this prospective cohort study is to investigate the role of Fluciclovine Positron Emission Tomography (PET) in patients with biochemical recurrence of prostate cancer (BCR) and a negative Prostate Specific Membrane Antigen (PSMA) PET, specifically, whether Fluciclovine PET can help detect local recurrence and whether the results of Fluciclovine PET can change management.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the detection rate of local recurrence of prostate cancer on Fluciclovine PET in patients with BCR and a negative or equivocal PSMA PET obtained within 30 days prior to the Fluciclovine PET.

SECONDARY OBJECTIVES:

I. To evaluate the correct localization rate of Fluciclovine PET in patients with positive scans.

II. To distinguish the detection rate by site of recurrence (local recurrence in the prostate bed, lymph node involvement, or distant metastatic disease), and stratify by PSA level at the time of the scan and tumor grade

III. To evaluate the change in management based on the results of Fluciclovine PET, relative to intended management based on the result of negative PSMA PET alone, prior to obtaining the Fluciclovine PET.

OUTLINE:

Patients will be imaged with Fluciclovine PET within 30 days of the negative or equivocal PSMA scan.

A short questionnaire inquiring about the intended management will be sent to the referring physician at two timepoints: 1) the first is at the time of screening, prior to the Fluciclovine PET; and 2) the second is after the availability of the results of Fluciclovine PET.

Change in intended management will be recorded. Participants will be followed for 6 months and will be managed by their treating physician as per standard-of-care.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Participant or legally authorized representative (LAR) must provide written informed consent before any study-specific procedures or interventions are performed.
* Patients with suspected BCR of prostate cancer after initial treatment, and a negative or equivocal PSMA PET, regardless of the findings on conventional imaging. Initial treatment may include prostatectomy and/or radiation therapy.
* PSA of 0.2 ng/mL or higher within 45 days of the scan.

Exclusion Criteria:

* Uncontrolled serious infection.
* Intercurrent illness or condition that would limit compliance with study requirements.
* Patients who have started any cancer treatment (systemic or radiation therapy) or who have started any supplements or herbal medications intended to treat cancer between the PSMA PET and Axumin PET/CT scans.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with BCR and a positive Fluciclovine PET performed within 30 days after a negative or equivocal PSMA PET | During PET scan procedure

SECONDARY OUTCOMES:
Correct localization rate (CLR) of Fluciclovine PET in patients with positive scans. | During PET scan procedure
  The CLR of Fluciclovine PET will be determined by the following formula: true positive/(true positive + false positive). This will be evaluated by patient, and only for patients in whom the standard-of-reference is available for analysis. Standard of reference, the combination of:
  1. Pathology, if site of recurrence is biopsied
  2. Drop in PSA levels if the site of recurrence undergoes radiation therapy
  3. Imaging follow up confirming the suspicious finding as true positive.
Number of participants with positive Fluciclovine PET summarized by site of recurrence (local recurrence in the prostate bed, lymph node involvement, or distant metastatic disease), stratified by PSA level | During PET scan procedure
Change in management based on the results of Fluciclovine PET, relative to intended management based on the result of negative PSMA PET alone, prior to obtaining the Fluciclovine PET. | Enrollment up to 1 month after scan
  Questionnaire filled by the referring physician stating the intended management at 2 timepoints, before and after the Fluciclovine PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Mallak, M.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States